CLINICAL TRIAL: NCT02666976
Title: The Prospective Study on the Effect of Ilaprazole in Non-erosive Reflux Disease Patients; Focused on Histologic Findings and Inflammatory Biomarker
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0110
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2016-01

CONDITIONS: Gastrointestinal Subepithelial Tumors
Keywords: Gastroesophageal reflux, proton pump inhibitors, ilaprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — ilaprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ilaprazole group (Experimental): ilaprazole 20mg once daily for 4 weeks.
  Interventions: Drug: Ilaprazole

INTERVENTIONS:
Drug: Ilaprazole — Patients who were diagnosed clinically as NERD and were treated with ilaprazole 20mg once daily for 4 weeks. Biopsies were obtained from 3cm above the EG junction before and after treatment. GERD Q questionnaire, histologic findings (basal cell hyperplasia, papillary elongation, dilated intercellular spaces, intraepithelial eosinophils and intraepithelial T lymphocyte) and inflammatory biomarkers (TNF-α, IL-8, IL-1β, TRPV1 and MCP-1) were accessed.

SUMMARY:
Non-erosive reflux disease (NERD) patients used to be less responsive to proton pump inhibitor (PPI)s as compared with patients with erosive esophagitis. The aim of this study is to objectively evaluate the effect of a new PPI, ilaprazole in NERD for adjusting the focus of symptom score, histopathologic findings and inflammatory biomarker.

A prospective study performed at single hospital enrolled 20 patients who were diagnosed clinically as NERD. Patients underwent EGD, a 24hr-combined multichannel intraluminal impedance and pH esophageal monitoring (MII-pH) and were treated with ilaprazole 20mg once daily for 4 weeks. Biopsies were obtained from 3cm above the EG junction before and after treatment. GERD Q questionnaire, histologic findings (basal cell hyperplasia, papillary elongation, dilated intercellular spaces, intraepithelial eosinophils and intraepithelial T lymphocyte) and inflammatory biomarkers (TNF-α, IL-8, IL-1β, TRPV1 and MCP-1) will be accessed.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years old and younger than 80 years old
* Patients with typical reflux symptoms at least 2days per week (or GERD Q score ≥ 8 )
* No erosion at GE junction through endoscopy
* Patients that can perform a 24 hr - combined multichannel intraluminal impedance and pH esophageal monitoring prior to this study.

Exclusion Criteria:

* included prior history of documented intolerance of ilaprazole or similar PPIs, or
* unsuspected alarm symptoms such as weight loss, hematemesis, hematochezia, jaundice or other significant illness like malignancy
* alcoholism or drug addiction
* uncontrolled diabetes, cerebrovascular accident or diseases needed an operation in the last 3 months before enrollment
* any previous esophageal surgery
* malignancy in gastrointestinal tract within 5years
* pregnant woman
* Zollinger-Ellison syndrome, Barrett's esophagus, primary esophageal motility abnormality, esophageal stricture, duodenal ulcer, gastric ulcer, pancreatitis, absorption disorder, severe cardiovascular disease, severe lung disease in the last 3 months before enrollment
* history of steadily taking medicine such as diazepam, quinidine, diphenylhydantoin, mephenytoin, warfarin, anticholinergic, prostaglandin analog, antineoplastic agent, salicylate, steroid, pro-motility drug, nonsteroidal anti-inflammatory drugs(NSAIDS)
* patients who were registered other exams within 28days
* patients who could not conduct sedated endoscopy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes of symptoms | 4 weeks
  All patients complete the GerdQ questionnaire before and after taking ilaprazole. It was utilized to assess improvement of symptoms after taking medicine.

SECONDARY OUTCOMES:
changes of histopathological findings | 4 weeks
  Changes of histopathological findings and inflammatory biomarkers will be assessed before and after treatment. Histologic findings include basal cell hyperplasia, papillary elongation, dilated intercellular spaces, intraepithelial eosinophils and intraepithelial T lymphocyte. Inflammatory biomarkers (TNF-α, IL-8, IL-1β, TRPV1 and MCP-1) were also accessed by RT-PCR.
changes of inflammatory biomarkers | 4 weeks
  Changes of histopathological findings and inflammatory biomarkers will be assessed before and after treatment. Histologic findings include basal cell hyperplasia, papillary elongation, dilated intercellular spaces, intraepithelial eosinophils and intraepithelial T lymphocyte. Inflammatory biomarkers (TNF-α, IL-8, IL-1β, TRPV1 and MCP-1) were also accessed by RT-PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No